CLINICAL TRIAL: NCT01727271
Title: An Open-Label, Pilot, Randomized, Multi-Center Study to Compare Efficacy and Safety of Tenofovir Monotherapy Alone With Tenofovir Monotherapy Followed by Concurrent Combination of Pegylated Interferon-Alpha-2b and Tenofovir or Tenofovir Monotherapy Followed by Sequential Therapy of Pegylated Interferon-Alpha-2b and Tenofovir in HBeAG-Positive Chronic Hepatitis B Patients With Raised ALT.
Brief Title: A Study to Compare Efficacy and Safety of Tenofovir Used Alone or in Combination With Pegylated Interferon Alpha-2b in Participants With Chronic Hepatitis B and Elevated Alanine Aminotransferase (MK-4031-384)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4031-384
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tenofovir Monotherapy (Active Comparator): Tenofovir 300 mg tablet, orally (PO) once daily for 8 weeks, then Tenofovir 300 mg tablet, PO, once daily for an additional 96 weeks (total treatment duration 104 weeks)
  Interventions: Drug: Tenofovir
- PegIFN-2b/Tenofovir Sequential Therapy (Experimental): Tenofovir 300 mg tablet, PO, once daily for 8 weeks, then PegIFN-2b, 1.5 mcg/kg subcutaneously (SC), once weekly, for 24 weeks, then Tenofovir 300 mg tablet, PO, once daily for 72 weeks (total treatment duration 104 weeks)
  Interventions: Drug: Tenofovir; Biological: Pegylated interferon alpha-2b
- Peg-IFN-2b + Tenofovir Combination Therapy (Experimental): Tenofovir 300 mg tablet, PO once daily for 8 weeks, then pegIFN-2b, 1.5 mcg/kg SC once weekly and tenofovir 300 mg tablet, PO, once daily for 24 weeks, and then tenofovir 300 mg tablet, PO, once daily for 72 weeks (total treatment duration 104 weeks)
  Interventions: Drug: Tenofovir; Biological: Pegylated interferon alpha-2b

INTERVENTIONS:
Drug: Tenofovir
  Other Names: Truvada
Biological: Pegylated interferon alpha-2b
  Other Names: SCH 054031; MK-4031
  Arms: Peg-IFN-2b + Tenofovir Combination Therapy; PegIFN-2b/Tenofovir Sequential Therapy

SUMMARY:
This study will compare monotherapy with tenofovir to sequential therapy with pegylated interferon alpha-2b (pegIFN-2b) followed by tenofovir, and to combination therapy with pegIFN-2b + tenofovir, in participants with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B and elevated alanine aminotransferase (ALT). All enrolled participants will be be administered tenofovir alone for 8 weeks and then will be randomly assigned to 1 of the 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (hepatitis B surface antigen [HBsAg]-positive for >6 months or evidence of chronic hepatitis B in liver biopsy)
* Elevated serum ALT level
* Liver biopsy or a non-invasive investigation within 12 months prior to randomization with Chronic Hepatitis B
* Treatment naïve or history of interferon for not more than 1 month, taken at least 6 months before enrollment
* Compensated liver disease

Exclusion Criteria:

* Known hypersensitivity to tenofovir, interferon alpha-2b, and/or any other component of the study products
* Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
* Need for prolonged or frequent use of systemic acyclovir or famciclovir
* Previously received lamivudine or an investigational anti-hepatitis B virus (HBV) nucleoside or nucleotide analog and were resistant to these drugs
* History of variceal bleeding or other GI bleeding due to portal hypertension, hepatic encephalopathy, spontaneous bacterial peritonitis, Grade III and IV esophageal varices unless banded or other clinical signs of hepatic decompensation
* History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC
* Need for potentially hepatotoxic drugs (e.g. dapsone, erythromycin, fluconazole, ketoconazole, rifampin, and anti-tuberculosis regimens) or nephrotoxic drugs (e.g. frequent nonsteroidal anti-inflammatories, aminoglycosides, amphotericin B, and foscarnet)
* One or more additional known primary or secondary causes of liver disease, other than hepatitis B
* History of clinical pancreatitis
* Pregnant or breastfeeding
* Female participants of childbearing potential and male participants must be willing to use acceptable method of birth control.
* Medical condition that requires frequent or prolonged use of systemic corticosteroids
* Use of warfarin or other anticoagulants during 30 days prior to screening or if expected to be needed during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who responded to treatment | Week 128
Number of participants experiencing adverse events (AEs) | Up to 128 weeks
Number of participants discontinuing study therapy due to AEs | Up to 104 weeks